CLINICAL TRIAL: NCT01977404
Title: Nutritional Evaluation of Patients With Congestive Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-NV-0484-CTIL
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Congestive Heart Failure
Keywords: Congestive heart failure; Energy expenditure; Body composition; Caloric intake
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study objective is to assess the nutritional status of Patients With Congestive Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure patients between tne ages 40 to 90,all stages of the disease.

Exclusion Criteria:

* non

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with congestive heart failure between the ages 40 to 90 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Professor, Principal Investigator — The Tel Aviv Sourasky medical center, Ichilov
Locations (1):
- Sourasky medical center (Ichilov), Tel Aviv, Israel